CLINICAL TRIAL: NCT01870960
Title: Maxillary Sinus Floor Augmentation With Bioss® and Enamel Matrix Derivative: Evaluation of Osteogenic Properties
Acronym: EMDOGAIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 13-PP-01
Record Dates: First submitted 2013-05-30; First posted 2013-06-06 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Patient Who is Requiring Bilateral Sinus Floor Elevation and Necessity of Dental Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- right control (Other): the patient is his own control The right side will be treated as normal while the left side will also receive the emdogaim
  Interventions: Other: 7 patients will be recuting to received EMDOGAIM in left side
- left control (Other): the patient is his own control The left side will be treated as normal while the right side will also receive the emdogaim
  Interventions: Other: 7 patients will be recuting to received EMDOGAIM in right side

INTERVENTIONS:
Other: 7 patients will be recuting to received EMDOGAIM in left side
  Arms: right control
Other: 7 patients will be recuting to received EMDOGAIM in right side
  Arms: left control

SUMMARY:
The main problem of using xenogenic bone in sinus floor elevation is the slow rate of absorption, which gives the percentages of vital bone low (20 to 30% depending on the study) in which the dental implant will be positioned However, osseointegration of the implant can be achieved only in vital bone. Enamel Matrix Derivative, through their angiogenic and osteogenic properties known, could promote bone healing during surgery sinus floor elevation by increasing the percentage of vital bone reformed, when added to xenografts.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 45 years, postmenopausal women (ie with amenorrhea for more than a year).
* Subject requiring bilateral sinus floor elevation, in order to place two implants in grafted side.
* patients smoking less than 10 cigarettes per day
* patients having read and understood the information note on the study and signed the informed consent form.
* patients affiliated to the social security system.

Exclusion Criteria:

* Patient with absolute contra-indication for dental surgery: valvular heart disease at risk of infectious endocarditis, recent myocardal (≤ 12 months), organ transplants, recent placement of a coronary stent (≤ 12 months), transient ischemic attacks recurrent, cardiovascular instability, uncontrolled epilepsy, rheumatic fever.
* Patient with metabolic bone disease (Paget's disease, osteomalacia, osteogenesis imperfecta)
* Patient with an ASA score ≥ 3.
* Patient with absolute contra-indication to dental surgery
* Patient with severe hematologic disease
* Patient with I or type II diabetes
* Patients with previous or current acute illness or severe chronic cardiovascular, renal, hepatic, gastrointestinal, allergic, endocrine, neuro-psychiatric, considered by the investigator to be incompatible with the conduct of the study.
* Patients treated with retinoids, oral bisphosphonates, oral anticoagulants or anticonvulsants.
* Patient have or have had cancer of the upper aerodigestive tract treated by radiotherapy.
* Patient taking a steroidal or non-steroidal anti-inflammatory, anti-cancer or immunosuppressive chemotherapy in the last 6 months.
* Patient monitoring considered difficult by the investigator.
* Patient with poor oral hygiene incompatible with oral surgery.
* Patients with periodontal disease unstabilized
* Patient with oral dermatitis or adverse occlusion.
* Patient with an acute or chronic infection of the surgical site (osteomyelitis).
* Patient with a known allergy to collagen
* Patient with autoimmune disease
* Patient with a linguistic or mental incapacity to understand information
* Patient younger than 45 years old
* Patient trust under curatorship or judicial protection
* Patients aged over 45 premenopausal.
* Patient participating in another clinical study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Percentage of vital bone obtained within the grafted site | evaluated six month after dental surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France